CLINICAL TRIAL: NCT04921683
Title: Biomarkers of Thalamic LIFUP in Chronic Disorders of Consciousness
Brief Title: The Use of LIFUP in Chronic Disorders of Consciousness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Casa Colina Hospital and Centers for Healthcare (Other)
Collaborators: University of California, Los Angeles (Other); Tiny Blue Dot Foundation (Other)
Responsible Party: Principal Investigator, Caroline Schnakers, Assistant Director of Research, Casa Colina Hospital and Centers for Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRB#21-000091
Record Dates: First submitted 2021-05-17; First posted 2021-06-10 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Disorder of Consciousness; Vegetative State; Minimally Conscious State; Minimally Conscious State Plus; Minimally Conscious State Minus; Traumatic Brain Injury; CVA (Cerebrovascular Accident); Anoxia, Brain; Thalamic Infarction; Coma; Prolonged
MeSH Terms: conditions — Consciousness Disorders; Persistent Vegetative State; Brain Injuries, Traumatic; Stroke; Hypoxia, Brain; Coma

STUDY DESIGN:
Intervention Model Description: A single group model is when a group of subjects is administered treatment/exposure to device. Then it is measured and observed using behavioral and diagnostic tools over a specified amount of time throughout the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Treatment LIFUP (Experimental): LIFUP will be performed at the bedside using frameless stereotaxy. Specifically, the LIFUP transducer will be fit to the patient's head employing adjustable straps, and will be positioned over the patient's left temporal bone to minimize bone absorption and refraction. Accurate aiming will be ensured using the Brain Sight neuronavigation device, customized for tracking our LIFUP transducer. Following LIFUP, the patient will undergo a second EEG session, except for the EEG cap being fit to the patient's head prior to the LIFUP session so that, as soon as LIFUP administration is complete, the EEG paradigm can be promptly administered. The patient will then be allowed to rest (~1h).The patient will then be administered a second dose of tracer in order to undergo a second PET measurement. Finally, at the end-of-day, the clinical coordinator will collect an Adverse Event Questionnaire and will fit the PSG device for night monitoring.
  Interventions: Device: BX Pulsar 1002 (LIFUP) Low intensity Focused Ultrasound Pulsation

INTERVENTIONS:
Device: BX Pulsar 1002 (LIFUP) Low intensity Focused Ultrasound Pulsation — Administration of LIFUP will be performed at the bedside using frameless stereotaxy. Specifically, the LIFUP transducer will be fit to the patient's head employing adjustable straps, and will be positioned over the patient's left temporal bone, over the "temporal window" in order to minimize bone absorption and refraction. Accurate aiming will be ensured employing the BrainSight neuronavigation device, customized for tracking our LIFUP transducer (total ~10 min). Once satisfactory aiming is achieved, the LIFUP exposure will be initiated employing the settings described previously (which meet the FDA safety limits: ISPPA <= 190W/cm2, ISPTA <= 0.72W/cm2). Accurate aiming will be monitored in real-time throughout exposure using the Brain Sight Neuronavigation interface.

SUMMARY:
When patients survive a severe brain injury but fail to fully recover, they often enter a Disorder of Consciousness (DoC) --that is, a set of related conditions of decreased awareness and arousal including the Vegetative State (VS) and the Minimally Conscious State (MCS). When these conditions become chronic, there are no approved treatments to help bolster any further recovery. In prior work, we have shown the clinical feasibility and potential of Low Intensity Focused Ultrasound Pulsation (LIFUP) as a remarkably safe form of non-invasive brain stimulation in these conditions.

DETAILED DESCRIPTION:
In the present study, we propose taking the "next step" to assess whether LIFUP can affect objective and validated markers of DoC patient impairment (in the direction of lesser impairment). Specifically, patients will be admitted at Casa Colina Hospital for a 10-day (in-patient) protocol, and two follow-up sessions, conducted remotely (e.g., over the phone) at 7 and 30-days post-discharge. The full length of the study is 40 days from admission. Over the admission period, patients will undergo multiple measurements of validated biomarkers, including behavioral testing, brain metabolism (using Positron Emission Tomography), and electroencephalography, before and after one session of LIFUP to thalamus.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of VS or MCS based on the CRS-R .
2. Chronic status:

   * 3 months post-injury for non-traumatic etiologies
   * 12 months post-injury for traumatic etiology
3. 18 years of age or older.
4. If on a psychotropic medication regimen, that regimen will be stable for at least 4 weeks prior to entry to the study and the patient will be willing to remain on a stable regimen during the protocol.

Exclusion Criteria:

1. History of neurological disorder (other than the brain injury).
2. Unsuitability to undergo Magnetic Resonance (MR) assessment (e.g., non-MR compatible implants).
3. Unsuitability to undergo LIFUP neuromodulation (e.g., presence of non-bone implant or absence of bone under the expected positioning of the device by the left temporal bone window).
4. Manifest continuous spontaneous movement (which would prevent imaging)
5. Participation in another concurrent clinical trial.
6. Having undergone PET, CT, or other exam involving the use of ionizing radiation in the 12 months prior to the date of scheduled admission to Casa Colina.
7. Dependence on ventilator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-04-14 (Actual)

PRIMARY OUTCOMES:
Coma Recovery Scale-Revised | Coma recovery scale-revised is completed at enrollment and twice a day on Day 1-10, except for Day 4. Maximum score is 23 with a minimum of 0. Higher scores mean better outcome.
  Change in maximum total and subscale scores.
Electroencephalography | The EEG will be conducted at Day 3, 4, 7 and 10 of the study.
  Change in fast to slow frequency power spectrum density and in P3b amplitude.
Positron Emission Tomography | This will be conducted on Day 4.
  Assess change in local standard uptake value (SUV) and global SUV.
Polysomnography | This will be conducted Day 1-10 of the study.
  Change in nightly average density of sleep-spindles and sleep structure.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Schnakers, PhD, Principal Investigator — Casa Colina Hospital and Centers for Healthcare; Martin Monti, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Casa Colina Hospital, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Adams JH, Graham DI, Jennett B. The neuropathology of the vegetative state after an acute brain insult. Brain. 2000 Jul;123 ( Pt 7):1327-38. doi: 10.1093/brain/123.7.1327. PMID 10869046
- [Result] Monti MM, Schnakers C, Korb AS, Bystritsky A, Vespa PM. Non-Invasive Ultrasonic Thalamic Stimulation in Disorders of Consciousness after Severe Brain Injury: A First-in-Man Report. Brain Stimul. 2016 Nov-Dec;9(6):940-941. doi: 10.1016/j.brs.2016.07.008. Epub 2016 Jul 22. No abstract available. PMID 27567470
- [Result] Monti MM. Cognition in the vegetative state. Annu Rev Clin Psychol. 2012;8:431-54. doi: 10.1146/annurev-clinpsy-032511-143050. Epub 2012 Jan 3. PMID 22224835
- [Result] Pasquinelli C, Hanson LG, Siebner HR, Lee HJ, Thielscher A. Safety of transcranial focused ultrasound stimulation: A systematic review of the state of knowledge from both human and animal studies. Brain Stimul. 2019 Nov-Dec;12(6):1367-1380. doi: 10.1016/j.brs.2019.07.024. Epub 2019 Jul 31. PMID 31401074
- [Result] Schnakers C, Monti MM. Disorders of consciousness after severe brain injury: therapeutic options. Curr Opin Neurol. 2017 Dec;30(6):573-579. doi: 10.1097/WCO.0000000000000495. PMID 28901969
- [Result] Yoo SS, Kim H, Min BK, Franck E, Park S. Transcranial focused ultrasound to the thalamus alters anesthesia time in rats. Neuroreport. 2011 Oct 26;22(15):783-7. doi: 10.1097/WNR.0b013e32834b2957. PMID 21876461